CLINICAL TRIAL: NCT00948701
Title: Community Volunteers Promoting Physical Activity Among Cancer Survivors
Acronym: MFT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Bernardine M. Pinto, Professor, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 206208; 1R01CA132854-01A1 (NIH)
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Exercise; Physical activity; Community volunteers; Peer mentors; Peer coaches; Social support
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phone-based PA program (RTR Plus) (Experimental): The PA intervention consists of PA counseling, matched to participants' motivational readiness, plus educational materials. RTR volunteers or "coaches" will be asked to contact participants by telephone once a week for 12 weeks. The purpose of these calls is to build a supportive relationship with the participant, monitor PA participation, identify any health concerns, assist the participant to identify relevant barriers to PA and help her to problem solve to overcome such barriers.
  Interventions: Behavioral: Moving Forward Together 2
- Standard RTR services (RTR) (Active Comparator): RTR volunteers will contact the participants in this group by telephone once a week, providing support and information integral to RTR. The volunteers will also review the educational materials sent to all participants receiving RTR services. This will allow the volunteers to build a relationship with the participants over 12 weeks and ensure that these participants receive a minimal intervention, reducing the risk of attrition at the 12-week assessment.
  Interventions: Behavioral: Moving Forward Together 2

INTERVENTIONS:
Behavioral: Moving Forward Together 2 — RTR volunteers from the ACS will be trained to offer a 12-week telephone-based PA program as a supplement to standard 12-week RTR services.
  Other Names: MFT2

SUMMARY:
Physical activity programs, when offered in research settings, have been shown to improve quality of life and reduce fatigue among breast cancer survivors. The investigators are training Reach to Recovery volunteers at the American Cancer Society (New England Division) to provide a 12-week telephone-based physical activity program (RTR Plus) for breast cancer survivors. The comparison group of survivors will receive Reach to Recovery services (RTR). Physical activity, fatigue and other outcomes will be examined among 108 breast cancer survivors at the start of the program, at 12 weeks and 24 weeks. If the physical activity program is found to be effective, there is a potential for dissemination among the 13,000 Reach to Recovery volunteers across the U.S.

DETAILED DESCRIPTION:
The current study, a randomized controlled trial, represents the next step in our efforts to extend the research on physical activity to the community setting; community volunteers will deliver the intervention, thereby making physical activity interventions much more accessible to survivors. In partnership with the National ACS office (Atlanta, GA) and the New England ACS Division, researchers at the Miriam Hospital will share their skills, experience and resources to examine the effects of training RTR volunteers to deliver brief physical activity counseling to breast cancer survivors. Fifteen to twenty RTR volunteers will be trained to offer a 12-week telephone-based PA program as a supplement to 12-week RTR services (RTR Plus) vs. delivering the standard 12-week RTR services (RTR) to 108 breast cancer survivors. Assessments of physical activity, fatigue and other outcomes will be completed at baseline, 12 weeks and 24 weeks. Data on side-effects of the intervention and costs of intervention delivery will be tracked. If the proposed randomized trial demonstrates positive effects, the results will be used to design and support a dissemination trial of the effects of physical activity promotion to enhance cancer recovery in a community setting.

ELIGIBILITY:
Inclusion criteria:

* Women aged 21 years or over with Stage 0-3 breast cancer will be eligible if they:

  * Are requesting Reach to Recovery services from the American Cancer Society.
  * Have been diagnosed in the past 5 years with Stage 0-3 breast cancer.
  * Are able to read and speak English.
  * Are ambulatory.
  * Are sedentary (i.e., do not meet recommendations for moderate-intensity PA [30 minutes/ day or more for at least 5 days/ week] or vigorous-intensity PA [20 minutes/day or more for at least 3 days/week].
  * Are able to walk unassisted.
  * Have access to a telephone.

Exclusion criteria:

* Women with:

  * More advanced disease (Stage 4).
  * Medical or psychiatric problems (e.g., substance abuse, coronary artery disease, peripheral vascular disease, diabetes, and orthopedic problems) that may interfere with protocol adherence will not be included.
* Participants will be asked to provide consent for medical chart review to extract disease and treatment variables. Eligible participants will obtain medical clearance from their physicians.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity - recorded via accelerometer and through interviewer-administered Seven Day Activity Recall (7 day PAR). | Baseline, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Fatigue - assessed with FACT-F | Baseline, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bernardine M. Pinto, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- Centers for Behavioral and Preventive Medicine, The Miriam Hospital, One Hoppin Street, Suite 314, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Pinto BM, Dunsiger SI, DeScenza VR, Stein K. Mediators of physical activity outcomes in a peer-led intervention for breast cancer survivors. Psychooncology. 2023 Apr;32(4):619-627. doi: 10.1002/pon.6107. Epub 2023 Jan 27. PMID 36683179